CLINICAL TRIAL: NCT01905228
Title: A Phase 1 Trial of CBL0137 in Patients With Metastatic or Unresectable Advanced Solid Neoplasm
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incuron (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: I137-101
Record Dates: First submitted 2013-07-09; First posted 2013-07-23 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors; Glioblastoma
Keywords: Metastatic Advance Solid Neoplasms; Unresectable Advance Solid Neoplasms
MeSH Terms: conditions — Glioblastoma | interventions — CBLC137

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CBL0137 (Experimental): * Dose Level 9: 150 mg/m2, IV
  * Dose Level 10: 180 mg/m2, IV
  * Dose Level 11: 240 mg/m2, IV
  * Dose Level 12: 320 mg/m2, IV
  * Dose Level 13: 400 mg/m2, IV
  * Dose Level 14: 540 mg/m2, IV
  * Dose Level 15: 700 mg/m2, IV
  * Dose Level 16: 920 mg/m2, IV
  * Dose Level 17: 1200 mg/m2, IV
  * Dose Level 18: 1600 mg/m2, IV
  * Dose Level 19: 2100 mg/m2, IV
  * Dose Level 20: 2700 mg/m2, IV
  Interventions: Drug: CBL0137

INTERVENTIONS:
Drug: CBL0137 — All doses are administered intravenously on Days 1, 8 and 15 of every 28 day cycle.
  Number of Cycles: 2 or until progression or unacceptable toxicity develops
  Other Names: Curaxin

SUMMARY:
This is an open-label, multi-center, sequential groups, dose-escalation study of CBL0137 administered intravenously in participants with metastatic or unresectable advanced solid malignancies.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the maximally tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of CBL0137. The secondary objectives are to describe the dose-limiting toxicity (DLT) and adverse event profile of CBL0137, to describe the pharmacokinetic profile of CBL0137, to document any objective responses to CBL0137. This is a study of CBL0137 with a standard "3+3" design. Escalation will proceed to the MTD based on DLT in the 1st cycle in 1 of 6 participants in a cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological or cytological evidence of a solid neoplasm
* Patients enrolled in the expansion cohort must have at least one measureable lesion as defined by the RECIST 1.1 criteria for patients with systemic tumors or the RANO criteria for patients with gliomas;
* Patients with a systemic tumor must:

  * have metastatic or unresectable advanced solid tumors that have recurred or progressed following standard therapy or
  * no longer be candidates for standard therapy or
  * have tumors for which there is no standard therapy
* Patients with a glioma must:

  * have Grade III (anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma) disease, Grade IV (glioblastoma) disease, or diffuse intrinsic pontine glioma (DIPG) and;
  * have received prior therapy including radiation and drug therapy and;
  * have documented recurrent disease as defined in the RANO criteria;
* Patients must be ambulatory and have an ECOG Performance Score of 0 or 1;
* Patients or their legal representative must be able to provide written informed consent;
* Patients must have adequate bone marrow reserve as evidenced by:

  * White Blood Cell Count (WBC) > 3,000/µL
  * Absolute Neutrophil Count (ANC) > 1,500/µL
  * Platelet count (PLT) > 75,000/µL
  * Hemoglobin (HGB) > 8.0 gm/dL (patients may be transfused to achieve this HGB level);
* Patients must have adequate hepatic function as evidenced by:

  * Serum AST/ALT < 3X the upper limit of normal (ULN) for the reference lab (< 5X the ULN for patients with known hepatic metastases)
  * Serum bilirubin < 1.5 x the ULN for the reference lab;

Exclusion Criteria:

* Patients with active infection or with a fever > 38.50 C within 3 days of the first scheduled day of dosing;
* Patients with symptomatic CNS metastases who have not undergone surgery and/or radiotherapy and/or who are not neurologically stable;
* Patients with known hypersensitivity to any of the components of CBL0137;
* Patients who are receiving concurrent anticancer therapy;
* Patients receiving enzyme-inducing antiepileptic agents within 14 days prior to the start of study therapy;
* Males with mean QTcF values of > 450 msec and females with QTcF values of > 470 msec following 3 ECGs conducted 5 minutes apart from each other; patients who are known to have congenital prolonged QT syndromes; or patients who are on medications known to cause prolonged QT intervals on ECG;

Please speak with the PI for the complete Inclusion/Exclusion listing.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2019-05 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) | At the end of Cycle 1 (each cycle is 28 days)
  MTD is defined as dose level at which ≥6 participants have been treated and which is associated with a first-cycle DLT in ≤17% of the participants. Selection of RP2D from within the tolerated dose range will be based on evaluation of short- and long-term safety information together with findings relating to compliance, pharmacokinetics, pharmacodynamics and antitumor activity.

CONTACTS AND LOCATIONS:
Overall Officials: John Sarantopoulos, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Renuka Iyer, MD, Principal Investigator — Roswell Park Cancer Institue; Afshin Dowlati, MD, Principal Investigator — University Hospital of Cleveland; Manmeet Ahluwalia, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - CTRC at The University of Texas Healh Science Center at San Antonio, San Antonio, Texas